CLINICAL TRIAL: NCT03676868
Title: Biology of Cerebral Arteriovenous Malformations : Study of the Link Between Blood Biomarkers and the Haemorrhagic Prognosis of Cerebral Arteriovenous Malformations
Brief Title: Biology of Cerebral Arteriovenous Malformations and Prognosis of Cerebral Arteriovenous Malformations
Acronym: BioMAV
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JDS_2018_6
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Arteriovenous Malformations; Ruptured or Unruptured Cerebral Arteriovenous Malformations
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The cerebral arteriovenous malformations correspond to the formation of an entanglement of morphologically abnormal vessels called nidus, which shunt the blood circulation directly from the arterial circulation to the venous circulation.

The cerebral arteriovenous malformations are an important cause of hemorrhagic stroke.

The hypothesis is that cerebral haemorrhage associated with a cerebral arteriovenous malformations would come from peri-nidal micro-vessels, in connection with infiltration of leucocytes and / or defective maintenance of microvascular integrity by platelets.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with a cerebral AVM for which an intervention (endovascular treatment or surgery) or only clinical monitoring
* Express consent to participate in the study

And

* children
* Free informed and express consent of both holders of the minor patient's parental authority, or, by way of derogation and only if the other holder of parental authority cannot give his or her consent within a time limit compatible with the methodological requirements specific to the conduct of the research with regard to its purposes, of one of the two holders of parental authority

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breast feeding woman

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a cerebral arterioveinus malformation for which an intervention (endovascular treatment or surgery) or only clinical monitoring is planned
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2028-11-19 (Estimated); Study Completion 2028-11-19 (Estimated)

PRIMARY OUTCOMES:
Associaton between dosage of endothelial marker and the arteriovenous malformation pronostic | 6 months
  associaton between dosage of endothelial marker in blood samples and correlation with clinical outcome
Associaton between dosage of platelet and the arteriovenous malformation pronostic | 6 months
  Dosage of platelet in blood samples and correlation with clinical outcome
Associaton between dosage of neutrophilic and the arteriovenous malformation pronostic | 6 months
  Dosage of neutrophilic in blood samples and correlation with clinical outcome
Associaton between neo-angiogenesis activation markers and the arteriovenous malformation pronostic | 6 months
  Dosage neo-angiogenesis activation markers in blood samples and correlation with clinical outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Rotschild, Paris, France